CLINICAL TRIAL: NCT04379089
Title: Neurologic Manifestations of COVID 19 in Children
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: University of Utah (Other); Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Ericka Fink, Associate Professor, Division of Pediatric Critical Care Medicine, University of Pittsburgh
Other Study IDs: STUDY20060012; STUDY20040154 (Other: University of Pittsburgh); STUDY20040278 (Other: University of Pittsburgh)
Record Dates: First submitted 2020-04-30; First posted 2020-05-07 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2023-01

CONDITIONS: COVID; Neurologic Manifestations
Keywords: child; neurocritical care; COVID-19; neurologic manifestations
MeSH Terms: conditions — Neurologic Manifestations; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children <18: Infants, children, and young adults age < 18 years
  Admitted to the hospital with confirmed or presumed COVID-19 infection (includes admissions to emergency, ward, intensive care etc.)
  Interventions: Other: Observational study only

INTERVENTIONS:
Other: Observational study only — No Intervention

SUMMARY:
The purpose of this study is to perform a secondary analysis of pre-existing de-identified limited datasets obtained from sites participating in Tier 1 (STUDY20040154: Neurologic Manifestations of COVID 19 in Children) and Tier 2 (STUDY20040278: Neuro COVID - Outcomes). The data will be used to determine the prevalence and severity of neurological symptoms among patients requiring critical care admission for confirmed or suspected novel coronavirus (COVID-19) and to determine the predictors for limitation of care in the study population, as well as, the prognosis of neurologically injured patients admitted to the ICU during the COVID-19 crisis.

This study is sponsored by the Pediatric Neurocritical Care Research Group (PNCRG) and sponsored and funded in part by the Neurocritical Care Society.

DETAILED DESCRIPTION:
Early reports of COVID-19 indicate that adults experience a variety of neurological symptoms and diagnoses in approximately 36% of patients, including headaches, seizures, coma, encephalitis, and cerebrovascular events including ischemic stroke, intracranial hemorrhage, and cerebral venous sinus thromboses. In children, recent evidence highlights acute and long-term neurological manifestations due to other viral illnesses including Guillain Barre syndrome and neonatal microcephaly with Zika virus, encephalitis with H1N1 influenza, and acute flaccid paralysis with enterovirus-68. However, COVID-19 reports in children published thus far lack detailed information on the frequency and outcomes of neurological findings.

COVID-19 cases are rapidly rising internationally, with experts forecasting subsequent global surges and continued activity. Thus, it is imperative to accurately document prevalence and outcomes of the neurological aspects of COVID-19 specifically in children. Such data will serve to alert clinicians and families about the possibility that children may present with neurologic rather than "classic" symptoms of COVID-19 who nevertheless would warrant testing, and that neurologic events can occur subsequent to the diagnosis that may impact long-term outcomes (e.g., cognitive, emotional, physical health). The investigators anticipate that improved knowledge about neurologic manifestations in children will bolster personalized treatment and rehabilitation strategies to optimize child outcomes and inform future interventional studies.

ELIGIBILITY:
Inclusion Criteria:

* Infants, children, and young adults age < 18 years
* Admitted to the hospital with confirmed or presumed COVID-19 infection (includes admissions to emergency, ward, intensive care etc.)

Exclusion Criteria:

* none

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants, children, and young adults age < 18 years
Sampling Method: Probability Sample
Enrollment: 3568 (Actual)
Dates: Start 2020-04-29 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Prevalence | 1 year
  Determine the prevalence of neurological manifestations and association with outcome in children with confirmed or presumed COVID-19 and/or MISC hospitalized between January 2020 and December 2021.
Child and family health functions | 1 month post discharge
  Measure child and family health functions and health-related quality of life (HRQOL) outcomes post discharge in children with confirmed or presumed COVID-19 and/or MISC diagnoses.

CONTACTS AND LOCATIONS:
Overall Officials: Ericka L Fink, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Fink EL, Alcamo AM, Lovett M, Hartman M, Williams C, Garcia A, Rasmussen L, Pal R, Drury K, MackDiaz E, Ferrazzano PA, Dervan L, Appavu B, Snooks K, Stulce C, Rubin P, Pate B, Toney N, Robertson CL, Wainwright MS, Roa JD, Schober ME, Slomine BS. Post-discharge outcomes of hospitalized children diagnosed with acute SARS-CoV-2 or MIS-C. Front Pediatr. 2024 Feb 12;12:1340385. doi: 10.3389/fped.2024.1340385. eCollection 2024. PMID 38410766